CLINICAL TRIAL: NCT03091842
Title: Taking AIM at Breast Cancer: Targeting Adiposity and Inflammation With Movement to Improve Prognosis in Breast Cancer Survivors
Brief Title: Exercise Intervention in Targeting Adiposity and Inflammation With Movement to Improve Prognosis in Breast Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1B-16-11; NCI-2017-00070 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1B-16-11 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Cancer Survivor; Central Obesity; Estrogen Receptor Positive; Postmenopausal; Progesterone Receptor Positive; Stage I Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage III Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Obesity, Abdominal; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (CARE program) (Experimental): Patients undergo supervised CARE program over 50 minutes comprising of warm up over 5 minutes, moderate to vigorous aerobic and resistance exercises over 40 minutes, and cool down over 5 minutes 3 days per week for 16 weeks.
  Interventions: Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Group II (TARE program) (Experimental): Patients undergo supervised TARE program over 80 minutes comprising of warm up over 5 minutes, aerobic exercise over 15 minutes, resistance exercise over 55 minutes, and cool down over 5 minutes 3 days per week for 16 weeks.
  Interventions: Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment
- Group III (home-based stretching program) (Active Comparator): Patients undergo home-based stretching program comprising of one set of 3-4 static stretching exercises held for 30 seconds 3 days per week for 16 weeks. Patients receive instructional DVD and booklet of the flexibility exercises. Patients also complete a weekly activity log. After completion of the stretching program, patients may optionally undergo the CARE program as in group I.
  Interventions: Behavioral: Exercise Intervention; Other: Informational Intervention; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Exercise Intervention — Undergo supervised CARE program
  Arms: Group I (CARE program)
Behavioral: Exercise Intervention — Undergo supervised TARE program
  Arms: Group II (TARE program)
Behavioral: Exercise Intervention — Undergo home-based stretching program
  Arms: Group III (home-based stretching program)
Other: Informational Intervention — Receive instructional DVD and booklet of the flexibility exercises
  Arms: Group III (home-based stretching program)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
  Arms: Group I (CARE program); Group III (home-based stretching program)

SUMMARY:
This randomized phase II trial studies how well exercise intervention works in targeting adiposity and inflammation with movement to improve prognosis in stage I-III breast cancer survivors. Different types of exercise may reduce inflammation in fat tissue and minimize the risk of cancer recurrence related to being overweight or obese.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effects of a 4-month circuit, interval-based aerobic and resistance exercise (CARE) intervention on obesity-associated chronic inflammation.

SECONDARY OBJECTIVES:

I. To determine the effects of a 4-month CARE intervention on sarcopenic obesity.

TERTIARY OBJECTIVES:

I. To determine the effects of a 4-month CARE intervention on breast cancer prognosis and assess whether reductions in chronic inflammation are associated with breast cancer prognosis.

OUTLINE: Patients are randomized to 1 of 3 groups.

GROUP I: Patients undergo supervised CARE program over 50 minutes comprising of warm up over 5 minutes, moderate to vigorous aerobic and resistance exercises over 40 minutes, and cool down over 5 minutes 3 days per week for 16 weeks.

GROUP II: Patients undergo supervised traditional aerobic and resistance exercise (TARE) program over 80 minutes comprising of warm up over 5 minutes, aerobic exercise over 15 minutes, resistance exercise over 55 minutes, and cool down over 5 minutes 3 days per week for 16 weeks.

GROUP III: Patients undergo home-based stretching program comprising of one set of 3-4 static stretching exercises held for 30 seconds 3 days per week for 16 weeks. Patients receive instructional digital video disc (DVD) and booklet of the flexibility exercises. Patients also complete a weekly activity log. After completion of the stretching program, patients may optionally undergo the CARE program as in group I.

After completion of study, patients are followed up at week 34, 8 and 12 months, and then every year for 8 years.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal (at time of diagnosis; including artificial menopause induced by previous hysterectomy) women newly diagnosed (stage I-III) breast cancer low grade disease positive for estrogen and progesterone receptors
* Are centrally obese with the following criteria (determined by study team at eligibility screening): body mass index (BMI) > 30 kg/m^2 (calculated using height and weight; an upper limit BMI will not be set; we will rely on obtaining physicians' clearance to assess full eligibility) or body fat > 30% (estimated by bioelectrical impedance), and waist circumference > 35 inches (in)
* Have undergone a lumpectomy or mastectomy
* Have received and completed neoadjuvant or adjuvant chemotherapy and/or radiation therapy within the past 12 months
* Speak English or Spanish
* Is in breast cancer remission with no detectable disease present
* Able to initiate a supervised exercise program (free from any cardiovascular, respiratory or musculoskeletal disease or joint problems that preclude moderate physical activity)
* Free from history of chronic disease including uncontrolled diabetes, hypertension or thyroid disease
* Have not experienced a weight reduction >= 10% within past 6 months
* Currently participate in less than 60 minutes of structured exercise/week
* No planned reconstructive surgery with flap repair during trial and follow-up period
* May use adjuvant endocrine therapy if use will be continued for duration of study intervention
* Does not smoke (no smoking during previous 12 months)
* Willing to travel to the exercise facility at University of Southern California (USC)

Exclusion Criteria:

* Patients with metastatic disease
* Is not centrally obese
* Has not completed surgery, chemotherapy, or radiation treatment associated with their diagnosis
* History of any musculoskeletal, cardiorespiratory or neurological diseases that preclude the participation in exercise
* Participates in more than 60 minutes of structured exercise/week
* Is planning reconstructive surgery with flap repair during trial and follow-up period
* Currently smokes
* Is unable to travel to the exercise facility at USC

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-29 (Estimated); Primary Completion 2024-07-29 (Estimated); Study Completion 2025-07-29 (Estimated)

PRIMARY OUTCOMES:
Reduction of adipose tissue inflammation assessed by measuring M1 and M2 adipose tissue macrophages, crown-like structures, and adipose tissue secretion levels of inflammatory cytokines secreted | Up to 16 weeks
  Analyses for each of the continuous outcomes will involve mixed effects linear regression models, to incorporate the repeatedly measured outcomes. Dependent variables will be the 2- and 4-month measurements of trial outcomes assessed during and at the end of the intervention period. Independent variables will include two indicator variables for treatment group (TARE, attention control) relative to CARE, the baseline value of the outcome, and an indicator variable for measurement time (2-month/4-month). The treatment group effect (2 degrees of freedom) will test for differences in TARE and/or attention control, relative to CARE on the 2- and 4-month outcomes.

SECONDARY OUTCOMES:
Distant DFS defined as events that are either lethal (death from any cause) or a direct threat to patient survival (distant recurrence or second primary invasive cancer) | Up to 8 years
  Kaplan-Meier estimates and log-rank tests will be used to estimate and initially test cumulative survival probabilities by treatment group. Cox proportional hazards models will be used to compare treatment groups (with 2 indicator variables for treatment group).
Overall survival | From randomization to death from any cause, assessed up to 8 years
  Kaplan-Meier estimates and log-rank tests will be used to estimate and initially test cumulative survival probabilities by treatment group. Cox proportional hazards models will be used to compare treatment groups (with 2 indicator variables for treatment group).
Recurrence-free interval defined as events directly attributable to the original breast cancer including invasive ipsilateral breast tumor recurrence; local, regional or distant recurrence; and death from breast cancer | Up to 8 years
  A competing risks analysis will be conducted, with death modeled as a competing event, using the Fine-Gray proportional hazards model. Analyses will be presented unadjusted, as well as adjusted for prognostic variables (age, estrogen receptor (ER)/HER2 status, tumor size, presence/number of positive nodes, and surgery (mastectomy vs. breast-sparing).
Sarcopenic obesity assessed using dual energy X-ray absorptiometry | Up to 8 months
  Analyses for each of the continuous outcomes will involve mixed effects linear regression models, to incorporate the repeatedly measured outcomes. Dependent variables will be the 2- and 4-month measurements of trial outcomes assessed during and at the end of the intervention period. Independent variables will include two indicator variables for treatment group (TARE, attention control) relative to CARE, the baseline value of the outcome, and an indicator variable for measurement time (2-month/4-month). The treatment group effect (2 degrees of freedom) will test for differences in TARE and/or attention control, relative to CARE on the 2- and 4-month outcomes.

OTHER OUTCOMES:
Disease free survival (DFS) | From randomization to documentation of disease recurrence or death from any cause, assessed up to 8 years
  Kaplan-Meier estimates and log-rank tests will be used to estimate and initially test cumulative survival probabilities by treatment group. Cox proportional hazards models will be used to compare treatment groups (with 2 indicator variables for treatment group). Ancillary analyses will assess associations of inflammation measures with DFS. Results will be presented as hazard ratios, with 95% confidence intervals. Unadjusted and adjusted survival curves will be presented by treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dieli-Conwright, PhD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Kang DW, Wilson RL, Gonzalo-Encabo P, Norris MK, Hans M, Tahbaz M, Dawson J, Nguyen D, Normann AJ, Yunker AG, Sami N, Uno H, Ligibel JA, Mittelman SD, Dieli-Conwright CM. Targeting Adiposity and Inflammation With Movement to Improve Prognosis in Breast Cancer Survivors (The AIM Trial): Rationale, Design, and Methods. Front Oncol. 2022 Jun 20;12:896995. doi: 10.3389/fonc.2022.896995. eCollection 2022. PMID 35795051